CLINICAL TRIAL: NCT00741156
Title: The Acute Effects of the Angiotensin-converting Enzyme Inhibitor Enalaprilat on Flow Distribution After the Bidirectional Cavopulmonary Connection
Brief Title: The Acute Effects of the Angiotensin-converting Enzyme Inhibitor Enalaprilat on Flow Distribution
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Kyong-Jin Lee, Staff Cardiologist, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1000012255
Record Dates: First submitted 2008-08-25; First posted 2008-08-26 (Estimated); Results first posted 2015-12-18 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-11

CONDITIONS: Hypertension; Congestive Cardiomyopathy
Keywords: pediatric; hypertension; congestive cardiomyopathy; angiotensin-converting enzyme inhibitor; cardiac catheterization
MeSH Terms: conditions — Hypertension; Cardiomyopathy, Dilated | interventions — Enalaprilat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Enalaprilat (Experimental): enalaprilat 0.005-0.01 mg/kg intravenous x 1 dose
  Interventions: Drug: Enalaprilat

INTERVENTIONS:
Drug: Enalaprilat — Enalaprilat will be administered intravenously i.v. 0.005 - 0.01 mg/kg i.v. over 1 minute
  Other Names: Vasotec

SUMMARY:
The primary objective of this study is to study the acute effects of angiotensin-converting enzyme inhibitor (ACEI) on systemic, pulmonary and cerebral blood flow in post bidirectional cavopulmonary connection (BCPC) patients.

DETAILED DESCRIPTION:
The intermediate stage of the bi-directional cavopulmonary connection (BCPC) in the management algorithm of single ventricle palliation is a unique and extraordinary physiologic condition. It places the superior vena caval blood flow into series with the lungs i.e. pulmonary blood flow is partially dependent on cerebral vascular flow and resistance. Differential reduction in the resistances of the systemic, cerebral and pulmonary vascular beds will result in re-equilibrium of relative blood flows which translate to alterations in arterial oxygen tension and perfusion pressure. This concept is demonstrated by the differential effects of carbon dioxide (CO2) and oxygen (O2). CO2 vasodilates and oxygen (O2) vasoconstricts the cerebral vascular bed; the opposite is true in the lungs. Furthermore, studies have demonstrated that arterial CO2 tension (PaCO2) at hypercarbic levels is favourable to normocarbia in increasing pulmonary, systemic and cerebral blood flows and reducing systemic vascular resistance in acute post BCPC patients.

Administration of angiotensin-converting enzyme inhibitor (ACEI) and other systemic vasodilator drugs are well established for treatment of patients with hypertension and congestive cardiomyopathy in both pediatric and adult populations. Favourable manipulation of the flow to the different vascular beds has been reported in children with significant intra-cardiac shunts in which pulmonary blood flow is decreased relative to the increase in systemic blood flow as a result of reduction of systemic vascular resistance.

Guided by similar principles, ACEI therapy is administered to patients with single ventricle physiology to redistribute relative blood flows across the pulmonary and systemic vascular beds. To date, there exists no study examining the hemodynamic effects of ACEI on relative blood flows in the setting of single ventricle physiology and in particular, no study demonstrates its benefits. The effects of ACEI are unknown on the equilibrium of relative cerebral, systemic and pulmonary blood flows in the post-BCPC state. A relative increase in systemic blood flow, as effected by ACEI, at the expense of cerebral blood flow may potentially adversely decrease pulmonary blood and ultimately reduce arterial oxygen tension. On the other hand, some data suggests that ACEI's improve cerebral autoregulation function; in which drop in blood pressure will signal a vasodilatory response in the cerebral vascular bed which may be particularly advantageous in BCPC patients.

Enalaprilat is the active diacid of the ACEI enalapril maleate. Doses of 0.01 to 0.06 mg/kg i.v. have been safely administered in pediatric studies. Onset of action is 15 minutes and duration of action is up to 12-24 hours. The pharmacokinetics of this drug are ideal for the purpose of this study. In our institution, all patients undergo routine cardiac catheterization after the BCPC procedure for hemodynamic assessment and angiography of cardiac structures to assess for eligibility for the Fontan operation.

ELIGIBILITY:
Inclusion Criteria:

* BCPC patients at time of routine pre-Fontan catheterization
* Patients between the ages of 2 months and 5 years old

Exclusion Criteria:

* Patients who have had ACEI therapy within 24 hours of the procedure

Ages: 2 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2008-07; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyong-Jin Lee, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Enalaprilat: Enalaprilat : Enalaprilat will be administered intravenously i.v. 0.01 mg/kg i.v. over 1 minute
Period: Overall Study
Arm/Group | Enalaprilat
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Enalaprilat
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 2.3 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — SEX WAS NOT IDENTIFIED
  Male | NA — SEX WAS NOT IDENTIFIED
Region of Enrollment [Number; unit: participants]
  Canada | 12

OUTCOME MEASURES:

1. Primary Outcome: Systemic, Pulmonary and Cerebral Blood Flow at Baseline and After Enalaprilat
Time Frame: Baseline and after enalaprilat
Measure: Median (Inter-Quartile Range); unit: l/min/m2
Groups:
- Systemic Blood Flow Baseline: Systemic blood flow in baseline condition
- Systemic Blood Flow After Enalaprilat: Systemic blood flow 20 minutes after enalaprilat
- Pulmonary Blood Flow Baseline: Pulmonary blood flow baseline condition
- Pulmonary Blood Flow After Enaliprilat: Pulmonary blood flow 20 minutes after enalaprilat
- Cerebral Blood Flow Baseline: Cerebral blood flow at baseline
- Cerebral Blood Flow After Enalaprilat: Cerebral blood flow 20 minutes after enalaprilat
Arm/Group | Systemic Blood Flow Baseline | Systemic Blood Flow After Enalaprilat | Pulmonary Blood Flow Baseline | Pulmonary Blood Flow After Enaliprilat | Cerebral Blood Flow Baseline | Cerebral Blood Flow After Enalaprilat
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12
l/min/m2 | 1.4 [0.9 to 1.8] | 1.8 [1.0 to 2.2] | 1.9 [1.8 to 2.9] | 1.9 [1.6 to 2.5] | 1.9 [1.6 to 2.9] | 1.8 [1.6 to 2.5]
Statistical Analysis 1: Comparison: Systemic Blood Flow Baseline vs Systemic Blood Flow After Enalaprilat; Test type: Superiority or Other; p = 0.09, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Systemic, Pulmonary and Cerebral Resistance at Baseline and After Enalaprilat
Description: Systemic, pulmonary and cerebral resistance is compared at baseline and after enalaprilat
Time Frame: Baseline and after enalaprilat
Measure: Median (Full Range); unit: Wood units per metre squared
Groups:
- Systemic Resistance at Baseline: systemic resistance in baseline condition
- Systemic Resistance After Enalaprilat: systemic resistance is measured after enalaprilat
- Pulmonary Resistance at Baseline: pulmonary resistance at baseline is measured
- Pulmonary Resistance After Enalaprilat: pulmonary resistance is measured after enalaprilat
- Cerebral Resistance at Baseline: cerebral resistance is measured in baseline condition
- Cerebral Resistance After Enalaprilat: cerebral resistance is measured after enalaprilat
Arm/Group | Systemic Resistance at Baseline | Systemic Resistance After Enalaprilat | Pulmonary Resistance at Baseline | Pulmonary Resistance After Enalaprilat | Cerebral Resistance at Baseline | Cerebral Resistance After Enalaprilat
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12
Wood units per metre squared | 40.94 [26.63 to 67.83] | 20.26 [16.5 to 28.16] | 2.87 [1.03 to 4.47] | 2.54 [0.49 to 4.76] | 24.07 [15.79 to 38.1] | 17.32 [13.57 to 21.79]

ADVERSE EVENTS:
Time Frame: 24 hours
Description: during cardiac catheterization monitoring period.
Arm/Group | Enalaprilat
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes